CLINICAL TRIAL: NCT04256187
Title: Pros and Cons of Botulinum Injection Treatment in Cerebral Palsy: A Qualitative Study Examining the Caregiver's Perspectives
Brief Title: Pros and Cons of Botulinum Injection Treatment in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020.114
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy; Botulinum Toxin
Keywords: botulinum toxin; cerebral palsy; experiences; spasticity; caregivers
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy group: Caregivers of children who treated with botulinum toxin.
  Interventions: Other: Qualitative interview

INTERVENTIONS:
Other: Qualitative interview — Qualitative interviews to sample the patient's feelings, experiences and thoughts risen by the treatments in the program.

SUMMARY:
The aim of this study is to quantitatively record the opinions regarding the pros and cons of this treatment of the caregivers of children with cerebral palsy who had botulinum toxin applied in investigators' clinic.

DETAILED DESCRIPTION:
Spasticity is defined as an increase in physiological resistance of the muscles associated with a lack of supraspinal inhibition against passive strain. It is a common and prohibitive problem associated with an increase in tendon reflex and tension reflex associated with upper motor neuron dysfunction. One of the most common problems in patients with CP.

Methods used in the treatment of spasticity; medical therapy, physical therapy, intrathecal baclofen pump, botulinum toxin injection, and orthopedic correction operations. However, botulinum toxin type-A (BTX-A) injections, which are applied to the muscles especially for localized spasticity, have become an effective adjuvant option that increases the effectiveness of classical methods and diversifies the treatment options.

BTX-A, which is basically a chemodenervation method; It is a treatment method that blocks the transmission of signal in the neuromuscular junction by preventing the release of acetylcholine vesicles into the presynaptic space. In spastic muscles, relaxation can be achieved by correct injection. Botulinum toxin type A has been shown to be an effective and safe treatment for children to reduce spasticity.

In Turkish society, there is no study evaluating the caregivers' experiences and opinions about botox treatments of patients with the diagnosis of cerebral palsy and limited studies in the literature are from countries with different sociodemographic features such as the United States and the United Kingdom. Although these patients have been receiving this treatment in investigators' center for years, there is no study in the literature that evaluates the plus and minus aspects of caregivers' experiences in this regard.

ELIGIBILITY:
Inclusion Criteria:

* To be the caregiver of a patient under 18 years old with cerebral palsy
* No attempt has been made to reduce spasticity such as botulinum toxin injection in the last 3 months.

Exclusion Criteria:

* Not knowing Turkish
* Refusing to participate in the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Caregivers of children who treated with botulinum toxin.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Experience of Botulinum toxin treatment | Day 0
  Qualitative interview performed at one occasion where the caregivers describes the experience about the their childrens' botulinum toxin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Evkaya, Res. Asst., Principal Investigator — Physiotherapy and Rehabilitation Department, Maltepe University; Ozge Kenis Coskun, Asts. Prof., Principal Investigator — Physical Medicine and Rehabilitation Department, Marmara University, Istanbul; Pemra Cobek Unalan, Prof, Principal Investigator — Family Medicine Department, Marmara University, Istanbul
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Barry MJ. Physical therapy interventions for patients with movement disorders due to cerebral palsy. J Child Neurol. 1996 Nov;11 Suppl 1:S51-60. doi: 10.1177/0883073896011001S08. PMID 8959462
- [Result] Corry IS, Cosgrove AP, Duffy CM, McNeill S, Taylor TC, Graham HK. Botulinum toxin A compared with stretching casts in the treatment of spastic equinus: a randomised prospective trial. J Pediatr Orthop. 1998 May-Jun;18(3):304-11. PMID 9600553
- [Result] Lundy C, Lumsden D, Fairhurst C. Treating complex movement disorders in children with cerebral palsy. Ulster Med J. 2009 Sep;78(3):157-63. No abstract available. PMID 19907680
- [Result] Im D, McDonald CM. New approaches to managing spasticity in children with cerebral palsy. West J Med. 1997 Apr;166(4):271. No abstract available. PMID 9168686
- [Result] Whelan MA, Delgado MR. Practice parameter: pharmacologic treatment of spasticity in children and adolescents with cerebral palsy (an evidence-based review): report of the quality standards subcommittee of the american academy of neurology and the practice committee of the child neurology society. Neurology. 2010 Aug 17;75(7):669. doi: 10.1212/WNL.0b013e3181ec670b. No abstract available. PMID 20713958
- [Derived] Karadag-Saygi E, Kenis-Coskun O, Unalan PC, Evkaya-Acar A, Giray E, Akgulle AH. Pros and cons of botulinum toxin injection therapy in cerebral palsy: A qualitative study exploring caregivers' perspective. Child Care Health Dev. 2022 Jan;48(1):150-158. doi: 10.1111/cch.12915. Epub 2021 Oct 21. PMID 34623695